CLINICAL TRIAL: NCT02065492
Title: Effect of L-type Calcium Channel Blocker (Amlodipine) on Myocardial Iron Deposition in Thalassemic Patients With Moderate to Severe Myocardial Iron Deposition: A Randomized Pilot Study
Brief Title: Amlodipine for Myocardial Iron in Thalassemia
Acronym: AMIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr Babar S Hasan, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AMIT
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Thalassemia
Keywords: Thalassemia; Amlodipine; Chelation; T2*; MRI; Myocardial Iron
MeSH Terms: conditions — Thalassemia | interventions — Deferoxamine; Amlodipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Chelation & Amlodipine (Experimental): This arm will receive both chelation and amlodipine.
  Amlodipine will be administered as a single daily dose. It will be administered at a dose of 0.1 mg/kg/day or maximum of 2.5 mg/day.
  Standard Chelation therapy will be administered either by subcutaneous infusion of Deferoxamine (3-5 days a week) or oral Deferasirox (daily) or combination of Deferoxamine and Deferiprone.
  The dosage will depend on individual requirement, as determined by the treating hematologist.
  Interventions: Drug: Standard Chelation; Drug: Amlodipine
- Standard Chelation (Active Comparator): Deferasirox or Deferoxamine or Deferiprone. Patients in this arm will be administered only standard chelation therapy,either by subcutaneous infusion of Chelation therapy of Deferoxamine (3-5 days a week) or oral Deferasirox (daily) or combination of Deferoxamine and Deferiprone.
  The dosage will depend on individual requirement, as determined by the treating hematologist.
  This will serve as the control arm of the study without any additional intervention.
  Interventions: Drug: Standard Chelation

INTERVENTIONS:
Drug: Standard Chelation — This will comprise of standard chelation drugs (Deferasirox or Deferoxamine or Combination of Deferoxamine and Deferiprone).The dosage and drug used will depend on ferritin levels and individual requirement, as determined by the treating hematologist and will be in accordance with the Iron chelation guidelines from Pakistan Thalassemia Society.
  Other Names: Asunra or Kelfer or Desferal
Drug: Amlodipine — doses of 0.2 to 0.25 mg/kg/day PO would be given during this trial
  Other Names: L-type calcium channel blocker
  Arms: Standard Chelation & Amlodipine

SUMMARY:
Children with thalassemia may have high iron levels after receiving blood transfusions. These high iron levels can have damaging effects on the body, especially the heart. Conventionally only chelation therapy was given for prevention of iron buildup in the heart. However, current research has shown that another drug, amlodipine, also helps to slow down the deposition of iron in the heart. This study is designed to see if patients receiving amlodipine along with their regular chelation therapy have a slower rate of iron buildup in the heart when compared with patients who are receiving chelation only.

DETAILED DESCRIPTION:
Null Hypothesis There is no difference between the efficacy of chelation plus amlodipine therapy and chelation therapy alone in retarding the rate of myocardial iron deposition in thalassemia patients with iron overload and a constant transfusion need.

Alternate Hypothesis Chelation plus amlodipine therapy is more efficacious than chelation therapy alone in retarding the rate of myocardial iron deposition in thalassemia patients with iron overload and a constant transfusion need.

The aim of the investigators study is to determine if amlodipine, an L-type specific calcium channel blocker, in addition to the standard aggressive chelation therapy, can retard the deposition of iron in the myocardium of thalassemia patients with significant myocardial iron load with or without cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged ≥ 6 and ≤ 20 years managed at AKUH for at least 1 year
* ≥ 10 blood transfusion in life time
* Transfusion need ≥ 180 ml/kg/year
* Serum ferritin ≥ 1000 ug/dl
* Patient deemed capable of receiving chelation therapy (by treating hematologist) either subcutaneous infusion of Deferoxamine (Desferal) (3-5 days a week) or oral deferasirox (daily) or Defeperione (oral) or a combination of Desferal and Defeperione.
* Patients who have been on a stable chelation regimen ≥ 6 months
* Completed and signed Informed consent/assent.

Exclusion Criteria:

* Patients with known hypersensitivity to amlodipine.
* Patients with known sinoatrial nodal disease or aortic stenosis.
* Patients with known severe myocardial dysfunction, defined as A LV ejection fraction of ≤ 4 SD for age even without symptoms.
* Patients with known signs and symptoms of heart failure.
* Patients with a T2* value of < 4 ms on cardiac MRI.
* Patients with systolic blood pressures ≤ 2 SD for age (systemic hypotension) at the time of enrolment.
* Patients with previously diagnosed significant congenital heart diseases or acquired heart diseases other than thalassemia (as defined earlier).
* Patients with known contraindications to MRI (pacemakers, cerebral aneurysm metal clips, etc.)
* Patient with a known history of developing tetany after use of a calcium channel blocker
* Known pregnancy.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of amlodipine in retarding rate of myocardial iron deposition (Assessed by change in T2* times) | At baseline, and then at 6 months and 12 months from the start of the study
  Each patient will be randomized into either of two study arms: amlodipine plus chelation or chelation alone. All patients will undergo MRI and T2* imaging at baseline and then at 6 and 12 month follow-up visits. Efficacy of Amlodipine will be assessed using change in T2* times.

SECONDARY OUTCOMES:
Effect of amlodipine therapy on left ventricular size, systolic and diastolic function | At baseline and then at 6 months and 12 months from the start of the study
  Cardiac MRI and echocardiogram will be utilized to assess both systolic and diastolic function. Basic parameters such as left ventricular end diastolic volume, left ventricular systolic volume and the ejection fraction will be measured.
  Mitral Inflow Doppler as well as Tissue Doppler Imaging will be used to assess diastolic dysfunction.
  Conventional Pulsed Doppler Echocardiography will be utilized to derive the myocardial performance index (Tei Index) of each patient which will serve as a surrogate for systolic function.
  Peak global and segmental longitudinal left and right ventricular strain and strain rate will be calculated using speckle tracking by tracing images obtained from the apical 4-chamber view. Peak global and segmental right and left ventricular circumferential strain and strain rate will also be calculated from a parasternal, mid-cavity short axis view using speckle tracking also.
Efficacy of amlodipine in retarding liver iron content (mg/g) | At baseline and then at 6 months and 12 months from the start of the study
  Liver iron content will be measured using T2* imaging of the liver
Adverse effects of amlodipine therapy | At baseline and at 6 months and 12 months from the start of the study; at all visits to the Clinical Trial Unit pharmacy at the Aga Khan Hosptal for dispensing amlodipine and at all routine visits to the outpatient hematology clinic
  Data on adverse effects will be be collected using the adverse event form. The adverse effects anticipated include fatigue, nausea, edema, palpitations, flushing, headache, dizziness, blurred vision, somnolence, cough, hypertension and sinus bradycardia. Any other adverse event will also be reported. Adverse events that require only symptomatic management will be treated by the participant's primary hematologist. Adverse events that require hospitalization will also be managed by the participant's primary hematologist and the costs incurred will be covered by the research fund. Cardiovascular adverse events that require outpatient or inpatient management will be treated by the Principal Investigator and his cardiology team and all costs incurred will be covered by the research fund.

CONTACTS AND LOCATIONS:
Overall Officials: Babar Hasan, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597
- [Derived] Shakoor A, Zahoor M, Sadaf A, Alvi N, Fadoo Z, Rizvi A, Quadri F, Tipoo FA, Khurshid M, Sajjad Z, Colan S, Hasan BS. Effect of L-type calcium channel blocker (amlodipine) on myocardial iron deposition in patients with thalassaemia with moderate-to-severe myocardial iron deposition: protocol for a randomised, controlled trial. BMJ Open. 2014 Dec 8;4(12):e005360. doi: 10.1136/bmjopen-2014-005360. PMID 25492271